CLINICAL TRIAL: NCT02697981
Title: The Effect of Personalized Tailored Nutrition Counseling in Pregnant Women After Bariatric Surgery on Compliance and Nutritional Habits
Brief Title: Effect of Personalized Nutrition Counseling in Pregnant Women After Bariatric Surgery on Nutritional Status and Habits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0309-15 - RBM
Record Dates: First submitted 2016-02-03; First posted 2016-03-03 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Pregnancy
Keywords: sleeve gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Pregnant post bariatric surgery women will receive nutritional counseling from a specialist dietitian, to ensure a healthy balanced diet including adequate daily servings from all food groups, intake of essential nutrient during pregnancy such as iron and folic acid and limitation of high-sugar and fatty foods. Patients will also be advised concerning eating at scheduled times (e.g., 4-6 times daily), supplements, preference of water. Advice concerning healthy cooking methods will also be given, as well as advised to avoid soft drinks, drinking during meals, grazing and emotional eating, and fast foods. Subject of lifestyle in general - encouraged to incorporate suitable physical activity on most days, refraining from alcohol, and smoking. intervention: nutrition counseling
  Interventions: Behavioral: nutrition counseling
- control group (No Intervention): The control group is comprised of healthy pregnant women, of similar age, smoking behavior and background. No treatment will be given, just follow-up data collection.

INTERVENTIONS:
Behavioral: nutrition counseling — nutrition counseling and guidance.
  Other Names: follow-up
  Arms: intervention group

SUMMARY:
Background: Nutrition challenges follow bariatric surgery can intensify during pregnancy and may have a crucial effect on fetus. To the best of the investigators knowledge, the effect of nutritional counseling on improvement of maternal diet quality and eating habits among post- bariatric pregnant women has not been evaluated.

Objective: study aims to expand the existing limited knowledge in respect to post bariatric pregnant women's eating habits and quality of food intake, and to investigate the impact of nutrition counseling on these factors.

Design: This is a controlled clinical trial comparing post Laparoscopic sleeve gastrectomy (LSG) pregnant women who received nutritional counseling with age-matched control healthy pregnant women. Counseling will focus on improving quality of food consumption, eating habits and behavioral changes in order to improve the mother and the fetus' nutritional status Nutritional data and eating behavior will be obtained using 24 hours recall dietary records and the Family Eating and Activity Habit Questionnaire (FEAHQ).

DETAILED DESCRIPTION:
Introduction Pregnancy is a critical period that can determine health for years to come. Appropriate nutrition during pregnancy is key to improved survival and health status of offspring, and can prevent numerous disease states from infancy to adult life. In recent year, as obesity has become a rising problem, bariatric surgery is the only way for many women to increase the chances of fertility.

A possible adverse effect of this approach is high frequency of nutritional deficiencies reported among this population, which may be critical in cases of pregnancy.

The risk for sub-optimal nutritional status and consequently a potential risk of developing micro and macronutrients deficiencies in post bariatric pregnancies, are higher compared to non-surgical pregnant women, given the nutrition challenges brought about by the surgery such as food aversions, nausea, and vomiting beyond the increased nutritional requirements exist in healthy pregnancy. Furthermore, even without the existence of nutritional deficiencies, maternal diet quality has a critical effect on fetus. "Western" diet, high in fats and sugars, increased sympathetic nervous system activity and hyperactivity in rodent offspring that persisted into adulthood. However Investigation of diet quality during pregnancy among women with bariatric surgery has shown that 82% of women's diet quality needs improvement. Moreover, dietary modifications are mainly directed towards increased pollution safety rather than improving diet quality in order to improve the mother and the fetus' nutritional status.

To the best of the investigators knowledge, the effect of dietary counseling in post bariatric pregnant women has not been evaluated despite the findings about its importance and efficacy in studies on non-pregnant bariatric patient.

The aims of this study is to expand the existing limited knowledge in respect to post bariatric pregnant women's' eating habits and quality of food intake, and to investigate the impact of nutrition counseling on these factors, which to best of the investigators knowledge had never been published.

Intervention Patients from the intervention group will receive nutritional counseling from a specialist bariatric dietitian trained in pregnancy nutrition as well. The main goals are a healthy balanced diet including adequate daily servings from all food groups (dairy and egg, meat, vegetables, fruit, whole grain starches, and healthy fats), intake of essential nutrient during pregnancy such as iron and folic acid and limitation of high-sugar and fatty foods. In addition, the patients were advised concerning eating at scheduled times (e.g., 4-6 times daily), taking supplements, preference of water. Advice concerning healthy cooking methods will also be provided. Participants will be advised to avoid soft drinks, drinking during meals, grazing and emotional eating, as well as fast foods. Also the subject of lifestyle in general will be addressed, and participants will be encouraged to incorporate suitable physical activity on most days, refraining from alcohol, and smoking. As currently, no guidelines exist in the literature for nutrition or behavioral modifications for pregnancy after LSG, counseling is based on previously published literature for bariatric and healthy pregnancy nutrition separately.

Each participant will received 8 follow-up sessions for dietary counseling.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* Bariatric surgery
* Laparoscopic sleeve gastrectomy
* control group - healthy pregnant women

Exclusion Criteria:

* multiple pregnancy
* chronic diseases
* post 15 weeks pregnancy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Nutrient intake | at inclusion (Time 1),will be compared to recommendation for each individual
  24 hour dietary intake and a questionaires on eating habits.
Nutrient intake | gestational week 20 (time 2), will be compared to recommendation for each individual
  24 hour dietary intake and a questionaires on eating habits.
Nutrient intake | gestational week 30 (time 3), will be compared to recommendation for each individual
  24 hour dietary intake and a questionaires on eating habits.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Mc, Haifa, Israel

REFERENCES:
- [Background] Barker DJP. Sir Richard Doll Lecture. Developmental origins of chronic disease. Public Health. 2012 Mar;126(3):185-189. doi: 10.1016/j.puhe.2011.11.014. Epub 2012 Feb 10. PMID 22325676
- [Background] Bebber FE, Rizzolli J, Casagrande DS, Rodrigues MT, Padoin AV, Mottin CC, Repetto G. Pregnancy after bariatric surgery: 39 pregnancies follow-up in a multidisciplinary team. Obes Surg. 2011 Oct;21(10):1546-51. doi: 10.1007/s11695-010-0263-3. PMID 20820939
- [Background] Verger EO, Aron-Wisnewsky J, Dao MC, Kayser BD, Oppert JM, Bouillot JL, Torcivia A, Clement K. Micronutrient and Protein Deficiencies After Gastric Bypass and Sleeve Gastrectomy: a 1-year Follow-up. Obes Surg. 2016 Apr;26(4):785-96. doi: 10.1007/s11695-015-1803-7. PMID 26205215
- [Background] Guelinckx I, Devlieger R, Donceel P, Bel S, Pauwels S, Bogaerts A, Thijs I, Schurmans K, Deschilder P, Vansant G. Lifestyle after bariatric surgery: a multicenter, prospective cohort study in pregnant women. Obes Surg. 2012 Sep;22(9):1456-64. doi: 10.1007/s11695-012-0675-3. PMID 22644802
- [Background] Kafri N, Valfer R, Nativ O, Shiloni E, Hazzan D. Health behavior, food tolerance, and satisfaction after laparoscopic sleeve gastrectomy. Surg Obes Relat Dis. 2011 Jan-Feb;7(1):82-8. doi: 10.1016/j.soard.2010.09.016. Epub 2010 Oct 31. PMID 21126923
- [Background] Stein J, Stier C, Raab H, Weiner R. Review article: The nutritional and pharmacological consequences of obesity surgery. Aliment Pharmacol Ther. 2014 Sep;40(6):582-609. doi: 10.1111/apt.12872. Epub 2014 Jul 30. PMID 25078533
- [Background] Kaiser LL, Campbell CG; Academy Positions Committee Workgroup. Practice paper of the Academy of Nutrition and Dietetics abstract: nutrition and lifestyle for a healthy pregnancy outcome. J Acad Nutr Diet. 2014 Sep;114(9):1447. doi: 10.1016/j.jand.2014.07.001. PMID 25699300
- [Derived] Araki S, Shani Levi C, Abutbul Vered S, Solt I, Rozen GS. Pregnancy after bariatric surgery: Effects of personalized nutrition counseling on pregnancy outcomes. Clin Nutr. 2022 Feb;41(2):288-297. doi: 10.1016/j.clnu.2021.11.035. Epub 2021 Dec 2. PMID 34999322